CLINICAL TRIAL: NCT01113268
Title: Role of Candidate Genes/Signalling Pathways in the Progression Towards Heart Failure: Study in a Cohort of Patients With a First Myocardial Infarction (PREGICA Patient Collection : Genetic Predisposition to Heart Failure)
Brief Title: PREdisposition Genetical in Cardiac Insufficiency = Genetic Predisposition to Heart Failure
Acronym: PREGICA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P081116; 2010-A00156-33 (Other: IDRCB)
Record Dates: First submitted 2010-04-28; First posted 2010-04-29 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2022-06

CONDITIONS: ST Elevation (STEMI) Myocardial Infarction of Other Sites
Keywords: Patient collection; Cardiac remodelling; Echography; Magnetic Resonance Imaging; Gene polymorphisms; Biomarkers
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Cohort Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1:cohort (Other): Our main goal is to create a prospective cohort of 1500 patients with a first large myocardial infarction allowing us, in a second step, to identify susceptibility genes for the progression of patients towards chronic heart failure using a candidate gene/candidate pathway approach.
  Interventions: Other: Cohort

INTERVENTIONS:
Other: Cohort — Our main goal is to create a prospective cohort of 1500 patients with a first large myocardial infarction allowing us, in a second step, to identify susceptibility genes for the progression of patients towards chronic heart failure using a candidate gene/candidate pathway approach.

SUMMARY:
Our main goal is to create a prospective cohort of 1500 patients with a first large myocardial infarction allowing us, in a second step, to identify susceptibility genes for the progression of patients towards chronic heart failure using a candidate gene/candidate pathway approach. Our main hypothesis is that there is, for a given initial biomechanical stress (duration of the ischemic episode, size of the infarcted area, etc.), a variation in the individual susceptibility to develop left ventricular remodelling and to progress towards heart failure, and that this variation is linked to genetic variants between individuals.

DETAILED DESCRIPTION:
The research program comprises 4 phases: a selection phase at D0-D1, a pre-inclusion and an inclusion phase at D4±2, a visit at M6, and a 5 year follow up phase.

Visit at Day 0 - Day 1:

* The first 12-lead ECG, to be included in the observation book, is performed.
* The first blood sample is taken.

Visit at Day 4±2:

* The first transthoracic echocardiography is performed in all patients selected.
* In the presence of at least 3 akinetic LV segments at the transthoracic echocardiography, the patient is included.
* Demographic data, medical and surgical anteriority, detailed circumstances of occurrence of the MI and any other relevant information is obtained during an interview.
* The second 12-lead ECG is performed.
* The second blood sample is taken.
* The first MRI is performed (optional)

Visit at 6 months:

* The second transthoracic echocardiography is performed.
* The third 12-lead ECG is performed.
* The third blood sample is taken.
* A 24-hour Holter-ECG monitoring is performed (optional)
* The second MRI is performed (optional)

Five year follow up (phone contact until 7 years after inclusion):

Each patient included at day 4±2 will be contacted by phone 1, 2, 3, 4 and 5 years post-MI to obtain information regarding cardiovascular events and hospitalizations. If the patient cannot be contacted directly, we will try to contact a member of his/her family or his/her family physician.

ELIGIBILITY:
Inclusion Criteria:

*Selection criteria

Any patient hospitalised in the CCU of the participating centers:

* with a diagnosis of a first MI
* with ST segment elevation and/or Q wave at admission
* with troponin elevation
* seen within the first 24 hours after symptom onset
* aged between 18 and 80 years is selected.
* consent emergency clause: His/her informed consent is obtained and he/she signs the consent form or However, if a member of the patients' family is present, his/her consent must be obtained or no consent

  *Inclusion
* The first transthoracic echocardiography is performed at day 4±2 in all patients selected.
* In the presence of at least 3 akinetic LV segments at the transthoracic echocardiography, the patient is included.

Exclusion Criteria:

*Non-selection criteria:

* Informed consent not obtained.
* Patients with diagnosis of previous MI, hypertrophic or dilated cardiomyopathy, significant valvular heart disease, chronic atrial fibrillation, or pace maker or any permanently implanted device susceptible to interfere with LV remodelling.
* Patients with preexisting heart failure.
* Patients having undergone previous cardiac surgery.
* Patients having received chemotherapy susceptible to induce LV remodeling (anthracyclines).
* Patients with an associated short-time life-threatening disease.
* Patients with poor echogenicity.
* Patients without health insurance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2010-09-30 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Identification of patients with LV remodeling from those without remodelling | at day 4±2, at month 6
  Our main judgement criterion allowing to distinguish patients with LV remodeling from those without remodelling will be an increase in LV end-diastolic volume > 20% between day 4±2 and month 6 post-MI.

SECONDARY OUTCOMES:
Degree of LV remodelling | at month 6
  To evaluate the degree of LV remodelling (including ventricular arrhythmias) 6 months after a first ST-segment elevation myocardial infarction (STEMI) or Q-wave MI at the era of early revascularization.
Power of the mutations/ polymorphisms, biomarkers and other intermediate phenotypes identified in predicting cardiovascular events | years 3 to 7
  To evaluate the power of the mutations/ polymorphisms, biomarkers and other intermediate phenotypes identified in predicting cardiovascular events (rehospitalizations, reinfarction, occurrence of HF, transplantation, arrhythmias, death) in a 5-year patient follow-up (years 3 to 7).

CONTACTS AND LOCATIONS:
Overall Officials: Damien LOGEART, MD,PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pr Damien LOGEART, Paris, France

REFERENCES:
- [Derived] Masurkar N, Bouvet M, Logeart D, Jouve C, Drame F, Claude O, Roux M, Delacroix C, Bergerot D, Mercadier JJ, Sirol M, Gellen B, Livrozet M, Fayol A, Robidel E, Tregouet DA, Marazzi G, Sassoon D, Valente M, Hulot JS. Novel Cardiokine GDF3 Predicts Adverse Fibrotic Remodeling After Myocardial Infarction. Circulation. 2023 Feb 7;147(6):498-511. doi: 10.1161/CIRCULATIONAHA.121.056272. Epub 2022 Dec 9. PMID 36484260